CLINICAL TRIAL: NCT02436941
Title: Loma Linda University Medical Center Department of Radiation Medicine Patient Registry
Brief Title: Radiation Medicine Patient Registry, Loma Linda University Medical Center
Status: Enrolling by invitation | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: 53191
Record Dates: First submitted 2015-03-27; First posted 2015-05-07 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Protons; Photons

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 99 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Proton or Photon

SUMMARY:
For most cancers, long-term follow-up is the best measure of treatment effectiveness. The Department of Radiation Medicine at Loma Linda University Medical Center operates the James M. Slater, M.D., Proton Treatment and Research Center, the world's first hospital-based proton treatment facility. Patients have been treated at the Center since 1990. Radiation treatment has been expanded and refined since the Center's opening, and these changes have been based primarily on outcomes seen and evaluated in long-term follow-up.

The Radiation Medicine Patient Registry (a multi-year database), which began as an IRB-approved study in 2003, including detailed follow-up of study data collected from 1990 and onward, is designed to track all medical information from patients treated with proton therapy and/or conventional X-ray therapy at Loma Linda University Medical Center. Information gathered from patients treated years or even decades ago helps to determine the most effective use of proton and conventional radiation in caring for patients with cancers and other diseases.

DETAILED DESCRIPTION:
The patient registry will be posted to accomplish three objectives:

1. Perform retrospective research studies on diseases treated with proton therapy and conventional photon radiation.
2. Maintain regular and life-long contact with patients in order to obtain current identification, contact information, and self/parent-reported health status. This information is used to generate better understanding of treatment strategies and, in turn, increase benefits to patients.
3. Enable physicians to review of medical record information and so to identify subjects who may be eligible to participate in future research studies. This requires obtaining permission from registered participants that they may be contacted and asked if they are interested in participating in studies for which they may be eligible, as determined by their medical information contained in the registry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of benign or malignant tumors or other conditions deemed treatable by proton or conventional photon radiotherapy
* Willingness to sign an Informed Consent Document

Exclusion Criteria:

* There are no specific exclusion criteria, but patients who are unwilling to sign the ICD will not be included

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patients who have proton or conventional x-ray therapy
Sampling Method: Probability Sample
Enrollment: 75000 (Estimated)
Dates: Start 2003-10-20 (Actual); Primary Completion 2040-03 (Estimated); Study Completion 2050-10 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | One year
  Participants will be followed per protocol pre- during- and following treatment per protocol schedule

SECONDARY OUTCOMES:
Local recurrence | One year
  Participants will be followed per protocol pre- during- and following treatment per protocol schedule

OTHER OUTCOMES:
Number of patients with adverse events | One year
  Participants will be followed per protocol pre- during- and following treatment per protocol schedule
Overall survival & Long-term follow-up | One year
  Maintaining regular, lifetime contact with patients enables physicians to obtain current identification, contact information, and self/parent-reported health status that can, in turn, generate better understanding of treatment strategies and subsequent benefits to patients

CONTACTS AND LOCATIONS:
Overall Officials: Jerry D Slater, MD, Principal Investigator — Loma Linda University

REFERENCES:
- [Background] Slater JD. Development and operation of the Loma Linda University Medical Center proton facility. Technol Cancer Res Treat. 2007 Aug;6(4 Suppl):67-72. doi: 10.1177/15330346070060S411. PMID 17668955
- [Background] Slater JD. Clinical applications of proton radiation treatment at Loma Linda University: review of a fifteen-year experience. Technol Cancer Res Treat. 2006 Apr;5(2):81-9. doi: 10.1177/153303460600500202. PMID 16551128
- [Background] Bush DA, Do S, Lum S, Garberoglio C, Mirshahidi H, Patyal B, Grove R, Slater JD. Partial breast radiation therapy with proton beam: 5-year results with cosmetic outcomes. Int J Radiat Oncol Biol Phys. 2014 Nov 1;90(3):501-5. doi: 10.1016/j.ijrobp.2014.05.1308. Epub 2014 Jul 30. PMID 25084608
- [Background] Slater JM, Ling TC, Slater JD, Yang GY. Palliative radiation therapy for primary gastric melanoma. J Gastrointest Oncol. 2014 Feb;5(1):E22-6. doi: 10.3978/j.issn.2078-6891.2013.057. PMID 24490048
- [Background] Bush DA, Cheek G, Zaheer S, Wallen J, Mirshahidi H, Katerelos A, Grove R, Slater JD. High-dose hypofractionated proton beam radiation therapy is safe and effective for central and peripheral early-stage non-small cell lung cancer: results of a 12-year experience at Loma Linda University Medical Center. Int J Radiat Oncol Biol Phys. 2013 Aug 1;86(5):964-8. doi: 10.1016/j.ijrobp.2013.05.002. PMID 23845845
- [Background] Ling TC, Kang JI, Bush DA, Slater JD, Yang GY. Proton therapy for hepatocellular carcinoma. Chin J Cancer Res. 2012 Dec;24(4):361-7. doi: 10.3978/j.issn.1000-9604.2012.10.09. PMID 23359779
- [Background] Slater JD, Loredo LN, Chung A, Bush DA, Patyal B, Johnson WD, Hsu FP, Slater JM. Fractionated proton radiotherapy for benign cavernous sinus meningiomas. Int J Radiat Oncol Biol Phys. 2012 Aug 1;83(5):e633-7. doi: 10.1016/j.ijrobp.2012.01.079. PMID 22768992
- [Background] Bush DA, Slater JD, Garberoglio C, Do S, Lum S, Slater JM. Partial breast irradiation delivered with proton beam: results of a phase II trial. Clin Breast Cancer. 2011 Aug;11(4):241-5. doi: 10.1016/j.clbc.2011.03.023. Epub 2011 Jun 12. PMID 21729673
- [Background] Coen JJ, Bae K, Zietman AL, Patel B, Shipley WU, Slater JD, Rossi CJ. Acute and late toxicity after dose escalation to 82 GyE using conformal proton radiation for localized prostate cancer: initial report of American College of Radiology Phase II study 03-12. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):1005-9. doi: 10.1016/j.ijrobp.2010.06.047. Epub 2010 Oct 6. PMID 20932675
- [Background] Talcott JA, Rossi C, Shipley WU, Clark JA, Slater JD, Niemierko A, Zietman AL. Patient-reported long-term outcomes after conventional and high-dose combined proton and photon radiation for early prostate cancer. JAMA. 2010 Mar 17;303(11):1046-53. doi: 10.1001/jama.2010.287. PMID 20233822
- [Background] Bush DA, Kayali Z, Grove R, Slater JD. The safety and efficacy of high-dose proton beam radiotherapy for hepatocellular carcinoma: a phase 2 prospective trial. Cancer. 2011 Jul 1;117(13):3053-9. doi: 10.1002/cncr.25809. Epub 2011 Jan 24. PMID 21264826
- [Background] Slater JM, Slater JD, Wroe A. Proton radiation therapy in the hospital environment: conception, development, and operation of the initial hospital-based facility, Review of Accelerator Science and Technology, Vol 2 (2009), 35-62
- [Background] Slater JD. Twenty years of proton radiation therapy at Loma Linda University Medical Center. In U. Linz, editor. Ion beam therapy: fundamentals, technology, clinical applications. Berlin: Springer, 2012:581-595.
- [Background] Bush DA, Smith JC, Slater JD, Volk ML, Reeves ME, Cheng J, Grove R, de Vera ME. Randomized Clinical Trial Comparing Proton Beam Radiation Therapy with Transarterial Chemoembolization for Hepatocellular Carcinoma: Results of an Interim Analysis. Int J Radiat Oncol Biol Phys. 2016 May 1;95(1):477-482. doi: 10.1016/j.ijrobp.2016.02.027. Epub 2016 Feb 13. PMID 27084661
- [Background] Bush DA, Slater JD, Shin BB, Cheek G, Miller DW, Slater JM. Hypofractionated proton beam radiotherapy for stage I lung cancer. Chest. 2004 Oct;126(4):1198-203. doi: 10.1378/chest.126.4.1198. PMID 15486383
- [Background] Slater JD, Rossi CJ Jr, Yonemoto LT, Bush DA, Jabola BR, Levy RP, Grove RI, Preston W, Slater JM. Proton therapy for prostate cancer: the initial Loma Linda University experience. Int J Radiat Oncol Biol Phys. 2004 Jun 1;59(2):348-52. doi: 10.1016/j.ijrobp.2003.10.011. PMID 15145147
- [Background] Bush DA, McAllister CJ, Loredo LN, Johnson WD, Slater JM, Slater JD. Fractionated proton beam radiotherapy for acoustic neuroma. Neurosurgery. 2002 Feb;50(2):270-3; discussion 273-5. doi: 10.1097/00006123-200202000-00007. PMID 11844261
- [Background] Slater JD, Yonemoto LT, Mantik DW, Bush DA, Preston W, Grove RI, Miller DW, Slater JM. Proton radiation for treatment of cancer of the oropharynx: early experience at Loma Linda University Medical Center using a concomitant boost technique. Int J Radiat Oncol Biol Phys. 2005 Jun 1;62(2):494-500. doi: 10.1016/j.ijrobp.2004.09.064. PMID 15890592
- [Background] Bush DA, Hillebrand DJ, Slater JM, Slater JD. High-dose proton beam radiotherapy of hepatocellular carcinoma: preliminary results of a phase II trial. Gastroenterology. 2004 Nov;127(5 Suppl 1):S189-93. doi: 10.1053/j.gastro.2004.09.033. PMID 15508084
- [Background] Bush DA, Slater JD, Bonnet R, Cheek GA, Dunbar RD, Moyers M, Slater JM. Proton-beam radiotherapy for early-stage lung cancer. Chest. 1999 Nov;116(5):1313-9. doi: 10.1378/chest.116.5.1313. PMID 10559093
- [Background] Slater JD, Rossi CJ Jr, Yonemoto LT, Reyes-Molyneux NJ, Bush DA, Antoine JE, Miller DW, Teichman SL, Slater JM. Conformal proton therapy for early-stage prostate cancer. Urology. 1999 May;53(5):978-84. doi: 10.1016/s0090-4295(99)00014-x. PMID 10223493
- [Background] Slater JD, Yonemoto LT, Rossi CJ Jr, Reyes-Molyneux NJ, Bush DA, Antoine JE, Loredo LN, Schulte RW, Teichman SL, Slater JM. Conformal proton therapy for prostate carcinoma. Int J Radiat Oncol Biol Phys. 1998 Sep 1;42(2):299-304. doi: 10.1016/s0360-3016(98)00225-9. PMID 9788407